## **Informed consent 29/07/2019**

## to participate in "Sarcopenia in acute care patients: Protocol

## for the European Collaboration of Geriatric Surveys:

## Sarcopenia 9+ EAMA project"

| Mr. / Ms. |
|---|
| National Identity Card # |
| [ ] I have read the information page I was given. |
| [ ] I have been able to ask my questions about the study. |
| [ ] I have spoken with Dr* |
| [ ] I understand that my participation is voluntary. |
| [ ] I understand that I can withdraw from the study at any time I want, without having to give any reason and without causing any repercussions for my medical care or health care services. |
| [ ] I agree to participate in the study. |
| [ ] I agree to be contacted in the upcoming months/years for eventual follow-up. |
| [ ] I agree that my clinical reports will be checked in the upcoming months/years for |
| eventual follow-up. |
| Signed, Signed, Dr. |
| In, 20 |